CLINICAL TRIAL: NCT05621070
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Efficacy and Safety of JS002 as Monotherapy in Patients With Primary Hypercholesterolaemia and Mixed Dyslipidemia
Brief Title: Efficacy and Safety of JS002 as Monotherapy in Patients With Primary Hypercholesterolaemia and Mixed Dyslipidemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS002-007
Record Dates: First submitted 2022-11-14; First posted 2022-11-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Hypercholesterolaemia and Mixed Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JS002 150mg Q2W (Experimental): JS002 150mg Q2W SC for 52 weeks
  Interventions: Drug: JS002
- JS002 450mg Q4W (Placebo Comparator): JS002 450mg Q4W SC for 52 weeks
  Interventions: Drug: JS002
- Placebo Q2W (Placebo Comparator): Placebo Q2W SC for 12 weeks, then switch to JS002 150mg Q2W SC for 40 weeks
  Interventions: Drug: Placebo
- Placebo Q4W (Placebo Comparator): Placebo Q4W SC for 12 weeks, then switch to JS002 450mg Q4W SC for 40 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS002 — JS002 will be administered per auto-injector. Participants will receive JS002 every 2 weeks subcutaneously.
  Arms: JS002 150mg Q2W
Drug: JS002 — JS002 will be administered per auto-injector. Participants will receive JS002 every 4 weeks subcutaneously.
  Arms: JS002 450mg Q4W
Drug: Placebo — Placebo will be administered per auto-injector. Participants will receive placebo every 2 weeks subcutaneously.
  Arms: Placebo Q2W
Drug: Placebo — Placebo will be administered per auto-injector. Participants will receive placebo every 4 weeks subcutaneously.
  Arms: Placebo Q4W

SUMMARY:
JS002 is a recombinant humanized anti-PCSK9 monoclonal antibody. This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, PK/PD profile, immunogenicity as well as complete delivery of auto-injector by patients of JS002 as monotherapy in patients with primary hypercholesterolaemia and mixed dyslipidemia.

In this study, two dose cohorts(150 mg, 450 mg) are set up, and 582 subjects are planned to be enrolled (randomizedly assigned to JS002 or placebo 150/450 mg group in a 2:1:2:1 ratio).A screening period (≤6 weeks), a double-blind treatment period (12 weeks), an open-label treatment period (40 weeks), and a follow-up period (8 weeks) will be required.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age 18~80 years old
3. Subject who has not achieve LDL-C goal as categorized by their CV risk at screening
4. Fasting TG≤4.5mmol/L by central laboratory at screening
5. Statin intolerance subject must have a history of statin intolerance as evidenced

Exclusion Criteria:

1. History of hemorrhagic stroke
2. NYHA III or IV heart failure, or known LVEF< 30% within 1 year before randomization
3. Uncontrolled serious cardiac arrhythmia defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response, or supraventricular tachycardia that are not controlled by medications, within 90 days prior to randomization
4. Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke, deep vein thrombosis or pulmonary embolism within 90 days prior to randomization
5. Planned cardiac surgery or revascularization
6. Uncontrolled hypertension defined as sitting systolic blood pressure(SBP) > 160 mmHg or diastolic BP (DBP) > 100 mmHg
7. Type 1 diabetes, poorly controlled type 2 diabetes (HbA1c > 8%), newly diagnosed type 2 diabetes (within 90 days of randomization)
8. Others factors not suitable for participation judged by PI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-09-23 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in LDL-C at Week 12 | Baseline and week 12
  Percent Change From Baseline in LDL-C at Week 12 in statin intolerance subjects
Percent Change From Baseline in LDL-C at Week 12 | Baseline and week 12
  Percent Change From Baseline in LDL-C at Week 12 in ITT subjects

SECONDARY OUTCOMES:
Change From Baseline in LDL-C at Week 12 | Baseline and week 12
  Change From Baseline in LDL-C at Week 12 in statin intolerance and ITT subjects
Percent Change From Baseline in LDL-C at Week 24,52 | Baseline and week 24,52
  Percent Change From Baseline in LDL-C at Week 24,52 in statin intolerance and ITT subjects
Change From Baseline in LDL-C at Week 24,52 | Baseline and week 24,52
  Change From Baseline in LDL-C at Week 24,52 in statin intolerance and ITT subjects
Percent Change From Baseline in other lipid parameters such as non-HDL-C, ApoB, TC, et al. at Week 12, 24, 52 | Baseline and week 12, 24, 52
  Percent Change From Baseline in other lipid parameters at Week 12, 24, 52 in statin intolerance and ITT subjects
Percentage of Participants With LDL-C Less Than 1.8 mmol/L(70 mg/dL) | Baseline and week 12, 24, 52
  Percentage of Participants With LDL-C Less Than 1.8 mmol/L(70 mg/dL) at Week 12, 24, 52 in statin intolerance and ITT subjects
Percentage of Participants With Full Administration of JS002 | Baseline and week 12, 24, 52
  Percentage of Participants With Full Administration of JS002 at Weeks 12, 24, 52 in statin intolerance and ITT subjects

OTHER OUTCOMES:
Number of Participants with anti-drug antibodies (ADAs) | From baseline to week 60
  Serum samples were analyzed for ADA. Positive samples were subsequently tested for neutralizing antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shao C, Zhang S, Cheng Z, Yang K, Wang G, Shi X, Yang H, Ji Y, Li H, Zhang S, Ma J, Pei Z, Zhang Y, Li Y, Li L, Zheng Y, Shao C, Zhang M, Hao Y, Tang YD. Efficacy and safety of ongericimab in Chinese statin-intolerant patients with primary hypercholesterolemia or mixed dyslipidemia: a randomized, placebo-controlled phase 3 trial. Atherosclerosis. 2025 Aug;407:120408. doi: 10.1016/j.atherosclerosis.2025.120408. Epub 2025 Jun 16. PMID 40543299